CLINICAL TRIAL: NCT04368806
Title: A 48-Weeks, Phase 2b/3a, Double-Blind, Randomized, Placebo Controlled, Multi-center, Superiority Study to Evaluate the Efficacy and Safety of JointStem, Autologous Adipose Tissue Derived Mesenchymal Stem Cells in Patients Diagnosed as Knee Osteoarthritis
Brief Title: A Phase 2b/3a Study to Evaluate the Efficacy and Safety of JointStem in Patients Diagnosed as Knee Osteoarthritis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nature Cell Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JS-OAP3-US01
Record Dates: First submitted 2020-04-21; First posted 2020-04-30 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- JointStem (Experimental): Autologous Adipose tissue derived Mesenchymal Stem Cells(AdMSC)
  Interventions: Drug: JointStem
- Placebo (Placebo Comparator): Normal Saline with Autologous Serum
  Interventions: Other: Placebo Control

INTERVENTIONS:
Drug: JointStem — Autologous Adipose tissue derived Mesenchymal Stem Cells (AdMSC)
  Arms: JointStem
Other: Placebo Control — Normal Saline with autologous Serum
  Arms: Placebo

SUMMARY:
This study is a double-blind, randomized, placebo controlled, multi-center, superiority study to evaluate the efficacy and safety of JointStem, autologous adipose tissue derived mesenchymal stem cells (AdMSC), in patients diagnosed as knee osteoarthritis. Following a 2-week screening period, approximately 140 subjects will be randomly assigned into one of the following two arms in a 1:1 ratio (1 JointStem : 1 Placebo). After each subject completes 48-Weeks visit (Visit 8) and the data management team confirms all individual data have no issue, the individual database will be locked and the blinding will be open for the statistical analysis.

DETAILED DESCRIPTION:
Study Procedures:

* Visit 1 (Week -7) - Screening
* Visit 2 (Week -5) - Baseline and Randomization (Lipoaspiration)
* Visit 3 (Week 0) - Treatment (Intra-articular injection)
* Visit 4 (Week 4) - 4 weeks follow-up
* Visit 5 (Week 12) - 12 weeks follow-up
* Visit 6 (Week 24) - 24 weeks follow-up
* Visit 7 (Week 36) - 36 weeks follow-up
* Visit 8 (Week 48) - 48 weeks follow-up (End of Study)

ELIGIBILITY:
<Inclusion Criteria>

1. Male or female of any race, adult aged 18 years or older
2. Subject who had osteoarthritis of knee diagnosed (according to the clinical and American College of Rheumatology Criteria)
3. Subject who has ≥ 45 on WOMAC function score at Screening and Baseline
4. Subject who has knee pain ≥ 70 mm for the study knee out of 100 mm on VAS (Visual Analog Scale) at Screening and Baseline
5. Subject who has radiographic evidence of grade 3 osteoarthritis in the study knee based on the Kellgren and Lawrence radiographic criteria
6. Subject who has a varus angle of 5 degrees or less confirmed through radiography
7. Subjects whose knee pain persists for at least 12 weeks (about 3 months) prior to Screening and does not improve symptoms with non-operative treatment options
8. Subject who is willing to discontinue all pain medications for osteoarthritis except rescue medication (acetaminophen < 3.25 g per day) at least 72 hours prior to Screening and throughout the duration of study
9. Subject who is willing and able to give written informed consent for participation in the study

<Exclusion Criteria>

1. Subject who has Body Mass Index (BMI) > 35 kg/m2
2. Subject judged by the investigator to have a history of clinically significant disease(s) (i.e., uncontrolled comorbid disease, kidney diseases, liver diseases, endocrine diseases, etc., but not limited to these diseases) that may affect the patient's participation in the study.
3. Subject who has any of following clinically significant diseases:

   * Autoimmune diseases
   * Paget's disease, ochronosis, acromegaly, hemochromatosis, or Wilson's disease
   * Genetic diseases (hyperkinesia, collagen gene abnormality, etc.)
   * Inflammatory joint disorders (e.g., rheumatoid inflammation)
   * Infectious joint disorders (e.g., septic arthritis)
   * Other joint disorders (e.g., gout, recurrent pseudogout, articular fracture, primary osteochondrosis, villonodular synovitis)
4. Subject who has any history of cancer and/or currently receiving treatment for a current cancer diagnosis.
5. Subject who is positive in pathogenic test (HIV, viral hepatitis, or syphilis)
6. Subject who has heart diseases (myocardial infarction, coronary artery bypass graft surgery, arrhythmia, or other serious heart diseases) or has history of heart diseases within 6 months prior to Screening
7. Subject who has received any intra-articular therapy in any joint within 6 months prior to Screening, or surgery on the relevant knee including articular endoscopic procedures within 6 months prior to Screening
8. Subject who has history of prolotherapy, or platelet rich plasma injection within 6 months prior to Screening
9. Subject who has received long-acting hyaluronic acid injection (e.g., Synvisc-One®, etc.) within 6 months prior to Screening
10. Subject who has history of stem cell therapy
11. Subject who has significant lab abnormalities for the following parameters (If the value is within 10% of the listed laboratory exclusion criterion value and the value is considered not to be clinically significant by the investigator, the subject can be considered for enrollment):

    * Serum ALT and AST > 2 x upper limit of normal
    * Serum creatinine out of normal range
    * PT/INR out of normal range
    * Hemoglobin < 10 g/dL for female subject and hemoglobin < 11 g/dL for male subject
    * Platelets out of normal range
12. Subject for whom the investigator judges the lipoaspiration can cause any problem
13. Subject who has history of local anesthetic allergy
14. Subject who has taken anti-inflammatory drugs (prescription and non-prescription NSAIDs), symptomatic slow acting drugs (glucosamine, chondroitin sulfate, diacerhein etc.), or oral steroids (prednisone etc.) within 14 days prior to Screening (however, those who undergo a 14-day wash-out period can participate.)
15. Subject who is an active drug/alcohol abuser
16. Pregnant or breast-feeding women, or women or men who are not using appropriate method of contraception (appropriate method includes hormones, bilateral tubal ligation, and barrier method with spermicide, and intra-uterine device for women and vasectomy and barrier method with spermicide for men; subjects should agree to use appropriate method)
17. Subject who is enrolled in any other clinical trials within 3 months from screening
18. Subject who received the COVID-19 vaccines within 1 week from Visit 2 (Lipoaspiration, baseline)
19. Subject who the principal investigator considers inappropriate for the study due to any other reasons than those listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) function Score | Baseline and Week 48
  Change from baseline in WOMAC function score at Week 48
Visual Analog Scale (VAS) score | Baseline and Week 48
  Change from baseline on Visual Analog Scale (VAS) score at Week 48

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) subscale (Function) | Week 12, 24 and 36
  Change from baseline in WOMAC subscale (Function) score at Week 12, 24, and 36
Western Ontario and McMaster Universities Arthritis Index (WOMAC) subscale (Pain) | Week 12, 24, 36, and 48
  Change from baseline in WOMAC subscale (Pain) score at Week 12, 24, 36, and 48
Total Western Ontario and McMaster Universities Arthritis Index (WOMAC) score | Week 12, 24, 36, and 48
  Change from baseline in total WOMAC score at Week 12, 24, 36, and 48
Visual Analog Scale (VAS) score | Week 12, 24 and 36
  Change from baseline in VAS score at Week 12, 24 and 36
International Knee Documentation Committee (IKDC) score | Week 12, 24, 36, and 48
  Change from baseline in IKDC score at Week 12, 24, 36, and 48
36-Item Short Form health survey questionnaires (SF-36) score | Week12, 24, 36, and 48
  Change from baseline in SF-36 score at Week 12, 24, 36, and 48
Kellgren-Lawrence grade | Week 48
  Change from screening in Kellgren-Lawrence grade of knee osteoarthritis determined by X-ray at Week 48
Number and amount of rescue medication use | Week 12, 24, 36, and 48
  The number and amount of rescue medication use at Week 12, 24, 36, and 48

CONTACTS AND LOCATIONS:
Locations (9):
- United States (5):
  - TriWest Research Associates, El Cajon, California
  - BioSolutions Clinical Research Center, La Mesa, California
  - Neurovations Research, Napa, California
  - Newport Therapeutics, Newport Beach, California
  - Source Healthcare, Santa Monica, California
- South Korea (4):
  - Keimyung University Dongsan Hospital, Daegu, Korea
  - Kyung Hee University Medical Center, Seoul, Korea
  - Kyung Hee University Hospital At Gangdong, Seoul, Korea
  - Smg-Snu Boramae Medical Center, Seoul, Korea